CLINICAL TRIAL: NCT03152682
Title: A Multi-centre Randomized, Double-blind, Placebo-controlled, Crossover, Proof-of-concept Study to Evaluate the Efficacy and Safety of Good IdeaTM on Glucose Homeostasis in a Healthy Population
Brief Title: A Study Evaluating Good Idea on Glucose Homeostasis in a Healthy Population
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: DoubleGood AB (Industry)
Collaborators: KGK Science Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 17GGHD
Record Dates: First submitted 2017-05-09; First posted 2017-05-15 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Healthy
Keywords: glucose; glucose homeostasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Consume GoodIdea at Visit 2 and Placebo at Visit 3 (Experimental)
  Interventions: Dietary Supplement: GoodIdea; Other: Placebo
- Consume Placebo at Visit 2 and GoodIdea at Visit 3 (Experimental)
  Interventions: Dietary Supplement: GoodIdea; Other: Placebo

INTERVENTIONS:
Dietary Supplement: GoodIdea — Active product. Amount: 355mL. Consumed at a clinic visit over 14 minutes.
Other: Placebo — Non-active placebo product. Amount: 355mL. Consumed at a clinic visit over 14 minutes.

SUMMARY:
A crossover design to evaluate the safety and efficacy of GoodIdea TM (trademark) on glucose homeostasis in a healthy population. Eligible participants will be given either the GoodIdea drink or placebo and a standardized meal and will consume both in approximately 15 minutes. Blood will be drawn at several time points over a 3 hour period to determine the study objectives. After a 7-day washout, the participants will come back to the clinic and and complete the visit consuming the opposite product given at the previous visit. The primary objective is to see the difference of the two-hour iAUC for intravenous blood glucose between the active product (GoodIdea) and the placebo following a standardized meal.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 to 50 years of age
* BMI 25-29.9 (±0.5) kg/m²
* Female participant is not of child bearing potential, which is defined as females who have had a hysterectomy or oophorectomy, bilateral tubal ligation or are post-menopausal (natural or surgically with > 1 year since last menstruation) OR
* Females of childbearing potential who agree to use a medically approved method of birth control and have a negative urine pregnancy test result. Acceptable methods of birth control include:
* Hormonal contraceptives including oral contraceptives, hormone birth control patch (Ortho Evra), vaginal contraceptive ring (NuvaRing), injectable contraceptives (Depo-Provera, Lunelle), or hormone implant (Norplant System)
* Double-barrier method
* Intrauterine devices
* Non-heterosexual lifestyle or agrees to use contraception if planning on changing to heterosexual partner(s)
* Vasectomy of partner (shown successful as per appropriate follow-up)
* White North American (should include Hispanic, non-Hispanic, Aboriginal and Asian) or African American
* Stable body weight defined as no more than ± 3 kg change during the last 2 months
* Agree to maintain consistent dietary habits and physical activity levels for the duration of the study
* Self-perceived general good health as per the general health questionnaire
* Fasting blood glucose < 6.1 mmol/L at screening
* Healthy as determined by laboratory results and medical history
* Willingness to complete questionnaires, records, and diaries associated with the study and to complete all clinic visits
* Has given voluntary, written, informed consent to participate in the study

Exclusion Criteria:

* Women who are pregnant, breast feeding, or planning to become pregnant during the trial
* Any medical condition(s) or medication(s) known to significantly affect glucose metabolism. Significance to be assessed by the Qualified Investigator
* Has undergone procedures that requires cleansing of the bowel, such as colonoscopy or barium enema within three months prior to randomization
* Type I or Type II diabetes
* Use of over-the-counter medication or natural health products that affect glucose metabolism is prohibited within 2 weeks of enrollment and during this study
* Use of anti-biotics within 2 weeks of enrollment
* Use of probiotic supplements within 2 weeks of enrollment
* Use of cholesterol lowering medications
* Use of blood pressure medications
* Use of over-the-counter decongestants that contain ephedrine or pseudoephedrine within 2 weeks of enrollment
* Use of acute or over the counter medications within 72 h of test product consumption
* Use of Tricyclic antidepressants or any other medication that will modify bowel function
* Metabolic diseases and chronic gastrointestinal diseases (IBS, Crohns etc.)
* Allergy to test product or placebo ingredients
* Participants restricted to a vegetarian or vegan diet
* Intolerance to lactose or gluten
* Irregular dietary habits, including: intermittent fasting, regularly skipped meals, and individuals who do not typically eat breakfast
* Any form of acute infection within 2 weeks of enrollment
* Individuals who are immuno-compromised (HIV positive, on anti-rejection medication, rheumatoid arthritis)
* History of gastrointestinal dysfunction or surgery that may influence digestion or absorption
* History of blood/bleeding disorders
* Individuals who are averse to venous catheterization or capillary blood sampling
* Current diagnosis of cancer, except skin cancers completely excised with no chemotherapy or radiation with a follow up that is negative. Volunteers with cancer in full remission for more than five years after diagnosis are acceptable
* Individuals who have planned surgery during the course of the study
* Alcohol or drug abuse within the last 6 months
* Currently active smokers (tobacco products, and e-cigarettes) or smoking within the 6 months of enrollment
* Blood or plasma donation in the past 2 months
* Participants planning to donate blood during, or within 30 days following completion of the study
* Use of medical marijuana
* History of, or current, psychiatric disease
* Unstable medical conditions as determined by Qualified Investigator
* Clinically significant abnormal laboratory results at screening
* Participation in a clinical research trial within 30 days prior to randomization
* Individuals who are cognitively impaired and/or who are unable to give informed consent
* Any other condition which in the Qualified Investigator's opinion may adversely affect the individual's ability to complete the study or its measures or which may pose significant risk to the individual
* Medical or psychological condition that in the Qualified Investigator's opinion could interfere with study participation

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-04-22 (Actual); Primary Completion 2017-08-15 (Actual); Study Completion 2017-08-15 (Actual)

PRIMARY OUTCOMES:
The difference of the two-hour iAUC (0 - 120 min) for intravenous blood glucose between Good IdeaTM and the placebo following a standardized meal. | 0 - 120 minutes

SECONDARY OUTCOMES:
The difference of the two-hour iAUC (0 - 120 min) for capillary blood glucose between Good IdeaTM and the placebo following a standardized meal. | 0 -120 minutes
The difference in the two-hour Cmax, (0 - 120 min) of capillary glucose between Good IdeaTM and the placebo following a standardized meal. | 0 - 120 minutes
The difference in the two-hour Tmax (0 - 120 min) of capillary glucose between Good IdeaTM and the placebo following a standardized meal. | 0 - 120 minutes
The difference in the two-hour iAUC (0 - 120 min) intravenous insulin iAUC between Good IdeaTM and the placebo following a standardized meal. | 0 - 120 minutes
The difference in the two-hour Cmax (0 - 120 min) of intravenous glucose and insulin between Good IdeaTM and the placebo following a standardized meal. | 0 - 120 minutes
The difference in the two-hour Tmax (0 - 120 min) of intravenous glucose and insulin between Good IdeaTM and the placebo following a standardized meal. | 0 - 120 minutes
The difference in the three-hour iAUC (0 - 180 min) for intravenous blood glucose and insulin between Good IdeaTM and the placebo following a standardized meal. | 0 - 180 minutes
The difference in the three-hour Cmax (0 - 180 min) of intravenous glucose and insulin between Good IdeaTM and the placebo following a standardized meal. | 0 - 180 minutes
The difference in the three-hour Tmax (0 - 180 min) of intravenous glucose and insulin between Good IdeaTM and the placebo following a standardized meal. | 0 - 180 minutes
The difference in the three-hour iAUC (0 - 180 min) of capillary glucose between Good IdeaTM and the placebo following a standardized meal. | 0 - 180 minutes
The difference in the three-hour (0 - 180 min) Tmax of capillary glucose between Good IdeaTM and the placebo following a standardized meal. | 0 - 180 minutes
The difference in the three-hour (0 - 180 min) Cmax, of capillary glucose between Good IdeaTM and the placebo following a standardized meal. | 0 - 180 minutes
Eating patterns as assessed by a 3-day food record for the weeks prior to days 0 and 8. | 1 week each

OTHER OUTCOMES:
The effects of supplementation with Good IdeaTM on vital signs (blood pressure) compared to placebo | 180 minutes
The effects of supplementation with Good IdeaTM on vital signs (heart rate) compared to placebo | 180 minutes
The change in Hematology from screening to end-of-study between Good IdeaTM and the placebo | 21 - 42 days
The change in Clinical chemistry from screening to end-of-study between Good IdeaTM and the placebo | 21-42 days
Incidence of adverse events in the Good IdeaTM and placebo group over the course of the study. | 8-14 days

CONTACTS AND LOCATIONS:
Overall Officials: Tetyana Pelipyagina, MD, Principal Investigator — KGK Science Inc.
Locations (1):
- KGK Synergize Inc., London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ostman E, Samigullin A, Heyman-Linden L, Andersson K, Bjorck I, Oste R, Humpert PM. A novel nutritional supplement containing amino acids and chromium decreases postprandial glucose response in a randomized, double-blind, placebo-controlled study. PLoS One. 2020 Jun 24;15(6):e0234237. doi: 10.1371/journal.pone.0234237. eCollection 2020. PMID 32579549